CLINICAL TRIAL: NCT01084564
Title: Economic Evaluation of Heart Failure Management in Colombian Clinics
Acronym: EconoHeart
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-CCO-ATA-2007/1
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Heart Failure; Asthma
Keywords: Cost-effectiveness analysis; Colombia
MeSH Terms: conditions — Heart Failure; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: moderate to severe uncontrolled asthma

SUMMARY:
Cost effectiveness analysis of local management of patients diagnosed with heart failure disease compared with an ideal guideline-based management.

ELIGIBILITY:
Inclusion Criteria:

* Asthma moderate to severe.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to severe uncontrolled asthma.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To determine cost-effectiveness of Heart Failure management in 3 Heart-specialized clinics in Bogotá Colombia | 12 months
Incremental cost-effectiveness ratio from using Symbicort as symbicort as Maintenance and Reliever Therapy (SMART) when compared with its competitive alternatives

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Dennis, M.D., Study Director — Pontificia Universidad Javeriana; MARÍA XIMENA ROJAS, M.D., Principal Investigator — Pontificia Universidad Javeriana